CLINICAL TRIAL: NCT04443062
Title: Lutetium-177-PSMA-617 Radioligand Therapy in Oligo-metastatic Hormone Sensitive Prostate Cancer.
Brief Title: Lutetium-177-PSMA-617 in Oligo-metastatic Hormone Sensitive Prostate Cancer
Acronym: Bullseye
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Prostaatkankerstichting (Unknown); Advanced Accelerator Applications (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL72585.091.20
Record Dates: First submitted 2020-06-17; First posted 2020-06-23 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-09

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; Hormone sensitive; Oligometastases; 177Lu-PSMA; Metastases directed therapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Pluvicto

STUDY DESIGN:
Intervention Model Description: Randomized, two-arm, open label, multi-center, phase II study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional arm: 177Lu-PSMA radioligand therapy (Experimental): 2 (+2) cycles of 7.4 GBq 177Lu-PSMA 6 weeks in between
  Interventions: Drug: 177Lu-PSMA-617
- Standard of care (No Intervention): Deferred androgen deprivation therapy. However, the control arm can receive the study drug (177Lu-PSMA) in case of disease progression (defined in the study protocol).

INTERVENTIONS:
Drug: 177Lu-PSMA-617 — PSMA radioligand therapy
  Arms: Interventional arm: 177Lu-PSMA radioligand therapy

SUMMARY:
Radioligand therapy (RLT) using Lutetium-177 labelled PSMA is a promising new therapeutic approach to treat metastatic prostate cancer. This tumor-specific treatment is directed against prostate-specific membrane antigen (PSMA), which is overexpressed in prostate cancer cells. In the last few years, several lutetium-177 (177Lu, β emitter) labeled PSMA ligands have been developed and are currently applied to treat metastatic castrate resistant prostate cancer patients. To date, there are no prospective randomized studies published using this treatment in the hormone sensitive setting or in oligometastatic prostate cancer. Therefore, this study we will evaluate the effect of 177Lu-PSMA in patients with hormone sensitive oligo-metastatic prostate cancer.

DETAILED DESCRIPTION:
Prostate-specific membrane antigen (PSMA) radioligand therapy (RLT) is a promising new therapeutic approach to treat metastatic prostate cancer. This tumor-specific treatment is directed against PSMA, which is overexpressed in prostate cancer cells. In the last few years, several Lutetium-177 (177Lu, β emitter) labeled PSMA ligands have been developed and are currently applied in nuclear medicine departments worldwide to treat metastatic castrate resistant prostate cancer (mCRPC) patients.

A large retrospective study reported an overall biochemical response rate of 45% following multiple 177Lu-PSMA RLT cycles in mCRPC patients, while 40% of patients already responded after a single cycle. RLT with 177Lu-PSMA was generally well tolerated and 12% of the patients suffered grade 3 to 4 hematological toxicity. In addition, mild and often transient xerostomia occurred in 8%. A prospective study carried out in Australia confirmed these results recently. Based on these outcomes Endocyte (a Novartis company) is currently carrying out an international multicenter prospective registration study for end-stage mCRPC patients (NCT03511664).

Although these results are promising, it is noteworthy that most of the currently available data is retrospective and 177Lu-PSMA has only been evaluated in end stage prostate cancer patients to date. However, based on the mode of action, 177Lu-PSMA could also be effective in low volume disease because of the very high tumor uptake of radioligands in smaller lesions. Also, in a pilot study (NCT03828838) we were able to show that 177Lu-PSMA treatment is safe coupled with promising response rates. Hence, the present randomized trial to investigate the efficacy of 177Lu-PSMA in patients with oligo-metastatic (≤5 metastases) metastatic prostate cancer, prior to the hormone insensitive state. In this study, 58 patients will be included in a 1:1 ratio to receive either 177Lu-PSMA or the current standard of care (deferred androgen deprivation therapy).

At the end of the study period for answering the primary research question, patients randomized to the control arm are eligible to receive 177Lu-PSMA if they meet the end of the study period treatment (EOT 1) criteria and are willing to undergo 177Lu-PSMA.

EOT 1 is defined by:

* Clinical progression determined by the treating physician (e.g. increasing pain from metastases)
* A 100% increase in PSA after cycle one blood draw (BASELINE) during study. Exception: PSA increase in the first 12 weeks after the first treatment injection as was defined by the PCWG3 criteria.

ELIGIBILITY:
Inclusion Criteria:

* Histological proven adenocarcinoma of the prostate with sufficient archived tumor material. This material has to be archived till study closure.
* Biochemical recurrence (PSA > 1.0 µg/l).
* PSA-doubling time < 6 months. Serum PSA progression is defined as 2 consecutive rising PSA values measured at least 1 week apart. The minimal start value is 0.2 µg/l.
* 18F-PSMA-PET-CT positive metastases in bones and/or lymph nodes (N1/M1ab): ≥1, maximally 5 metastases.
* Local treatment for oligo-metastases with radiotherapy or surgery appears to be no option anymore (due to prior treatment or the location of the metastatic lesions or if the patient refuse these treatments).
* No prior hormonal therapy (including any androgen directed treatment such as finasteride, dutasteride, bicalutamide, apalutamide, abiraterone or enzalutamide) or taxane based chemotherapy (docetaxel or cabazitaxel); testosterone > 1.7 nmol/l.

Exception: local prostate cancer treated with local radiotherapy plus adjuvant ADT; these patients need to be stopped with ADT at least 6 months.

* A detectable lesion on the 18F-PSMA PET/CT with significant PSMA avidity, defined by a SUVmax > 15 (partial volume corrected).
* ECOG 0-1
* Patients must have a life expectancy >6 months.
* Laboratory values:

  * White blood cells > 3.0 x 109/l
  * Platelet count > 75 x 109/l
  * Hemoglobin > 6.2 mmol/l
  * ASAT, ALAT < 3 x ULN
  * MDRD-GFR ≥ 50 ml/min
* Signed informed consent.

Exclusion Criteria:

* A known subtype other than prostate adenocarcinoma.
* Previous PSMA based radioligand treatment.
* Visceral or brain metastases.
* Any medical condition present that in the opinion of the investigator will affect patients' clinical status when participating in this trial.
* Prior hip replacement surgery potentially influencing performance of PSMA PET/CT.
* Sjogren's syndrome
* A second active malignancy other than prostate cancer.
* Patients who are sexually active and not willing/able to use medically acceptable forms of barrier contraception.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 58 (Estimated)
Dates: Start 2020-07-20 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
To compare the fraction of patients that have disease progression (and meet EOT 1) criteria within 6 months in a group of patients that are treated with 177Lu-PSMA and a group that follows the current standard of care. | 30 weeks
  Disease progression (EOT 1) is defined by:
  * A 100% increase in PSA after cycle one blood draw (BASELINE) during study. Exception: PSA increase in the first 12 weeks after the first treatment injection as was defined by the PCWG3 criteria. Or;
  * Clinical progression determined by the treating physician (e.g. increasing pain from metastases).
A second primary aim is to compare the two arms for the time to disease progression and meeting EOT 1 criteria. | 30 weeks
  Disease progression (EOT 1) is defined by:
  * A 100% increase in PSA after cycle one blood draw (BASELINE) during study. Exception: PSA increase in the first 12 weeks after the first treatment injection as was defined by the PCWG3 criteria. Or;
  * Clinical progression determined by the treating physician (e.g. increasing pain from metastases).

SECONDARY OUTCOMES:
To evaluate the clinical efficacy of multiple doses 177Lu-PSMA radioligand therapy in patients with oligo-metastatic, hormone sensitive metastatic PCa by: | 30 weeks
  The change in PSA after 177Lu-PSMA and proportion of achieving a ≥ 50% decrease in PSA from baseline.
To evaluate the clinical efficacy of multiple doses 177Lu-PSMA radioligand therapy in patients with oligo-metastatic, hormone sensitive metastatic PCa by: | 30 weeks
  The changes in uptake (SUVmax) of 18F-PSMA PET/CT before and 6 months after 177Lu-PSMA.
To evaluate the clinical efficacy of multiple doses 177Lu-PSMA radioligand therapy in patients with oligo-metastatic, hormone sensitive metastatic PCa by: | 30 weeks
  The size of soft tissue metastases on 18F-PSMA PET/CT and (whole body) MRI after 177Lu-PSMA.
Progression free survival defined as from the time from inclusion to date of evidence of clinical progression, death from any cause, PSA progression, or radiographic progression. | 30 weeks
  Clinical progression is defined by the treating physician (e.g. increasing pain from metastases). PSA progression is defined as a ≥ 25% increase in PSA from nadir, with a minimum PSA of >0,5 µg/l and which is confirmed by a second value ≥ 3 weeks later (i.e. confirmed rising trend). Within the first 12 weeks after treatment administration PSA increases will be ignored in the absence of other evidence of disease progression due to the flare phenomenon. If no decline occurs, date of ≥ 25% increase will be recorded. Radiographic progression is defined by the amount and size of the lesions. Where applicable PCWG3 and RECIST v1.1 criteria will be followed.
Time till initiation of ADT in patients receiving 177Lu-PSMA. ADT free survival is defined by the date any ADT (e.g. bicalutamide, LHRH, enzalutamide, abiraterone, etc.) is started or death related to PCa. | 30 weeks
To evaluate the tolerability and toxicity of 177Lu-PSMA defined by NCI Common Terminology Criteria for Adverse Events v5.0. | 30 weeks
To evaluate the quality of life before and up to 6 months after 177Lu-PSMA RLT. | 30 weeks
  The following questionnaires will be used: EORTC QLQ-C30, QLQ-PR25 & xerostomia inventory.

CONTACTS AND LOCATIONS:
Overall Officials: James Nagarajah, Prof., Principal Investigator — Radboud University Medical Center
Locations (4):
- German Oncology Center, Limassol, Cyprus
- Netherlands (3):
  - Amsterdam UMC, Amsterdam
  - University Medical Center Groningen, Groningen
  - Radboud University, Nijmegen

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rahbar K, Ahmadzadehfar H, Kratochwil C, Haberkorn U, Schafers M, Essler M, Baum RP, Kulkarni HR, Schmidt M, Drzezga A, Bartenstein P, Pfestroff A, Luster M, Lutzen U, Marx M, Prasad V, Brenner W, Heinzel A, Mottaghy FM, Ruf J, Meyer PT, Heuschkel M, Eveslage M, Bogemann M, Fendler WP, Krause BJ. German Multicenter Study Investigating 177Lu-PSMA-617 Radioligand Therapy in Advanced Prostate Cancer Patients. J Nucl Med. 2017 Jan;58(1):85-90. doi: 10.2967/jnumed.116.183194. Epub 2016 Oct 20. PMID 27765862
- [Background] Hofman MS, Violet J, Hicks RJ, Ferdinandus J, Thang SP, Akhurst T, Iravani A, Kong G, Ravi Kumar A, Murphy DG, Eu P, Jackson P, Scalzo M, Williams SG, Sandhu S. [177Lu]-PSMA-617 radionuclide treatment in patients with metastatic castration-resistant prostate cancer (LuPSMA trial): a single-centre, single-arm, phase 2 study. Lancet Oncol. 2018 Jun;19(6):825-833. doi: 10.1016/S1470-2045(18)30198-0. Epub 2018 May 8. PMID 29752180
- [Derived] Prive BM, Janssen MJR, van Oort IM, Muselaers CHJ, Jonker MA, van Gemert WA, de Groot M, Westdorp H, Mehra N, Verzijlbergen JF, Scheenen TWJ, Zamecnik P, Barentsz JO, Gotthardt M, Noordzij W, Vogel WV, Bergman AM, van der Poel HG, Vis AN, Oprea-Lager DE, Gerritsen WR, Witjes JA, Nagarajah J. Update to a randomized controlled trial of lutetium-177-PSMA in Oligo-metastatic hormone-sensitive prostate cancer: the BULLSEYE trial. Trials. 2021 Nov 4;22(1):768. doi: 10.1186/s13063-021-05733-4. PMID 34736509
- [Derived] Prive BM, Janssen MJR, van Oort IM, Muselaers CHJ, Jonker MA, de Groot M, Mehra N, Verzijlbergen JF, Scheenen TWJ, Zamecnik P, Barentsz JO, Gotthardt M, Noordzij W, Vogel WV, Bergman AM, van der Poel HG, Vis AN, Oprea-Lager DE, Gerritsen WR, Witjes JA, Nagarajah J. Lutetium-177-PSMA-I&T as metastases directed therapy in oligometastatic hormone sensitive prostate cancer, a randomized controlled trial. BMC Cancer. 2020 Sep 14;20(1):884. doi: 10.1186/s12885-020-07386-z. PMID 32928177